CLINICAL TRIAL: NCT02647229
Title: Measuring the Effectiveness and Utility of Colonic Irrigation for Bowel Preparation in Patients Undergoing Screening or Surveillance Colonoscopy
Brief Title: Colonic Irrigation for Colonoscopy Preparation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-01351
Record Dates: First submitted 2015-12-22; First posted 2016-01-06 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isosmotic bowel cleansing preparation (Active Comparator): Isosmotic solution ingested prior to colonoscopy
  Interventions: Other: Isosmotic bowel cleansing preparation
- Colonic Hyrdrotherapy (Active Comparator): Colonic hydrotherapy is an FDA approved method of colon cleansing using constant warm water lavage with a contained temperature and pressure controlled device administered by a trained technician.2 There
  Interventions: Other: Colonic Hyrdrotherapy

INTERVENTIONS:
Other: Isosmotic bowel cleansing preparation — Isosmotic Preps contain polyethylene glycol (PEG) and are osmotically balanced, high-volume, nonabsorbable, and nonfermentable electrolyte solutions.
  Arms: Isosmotic bowel cleansing preparation
Other: Colonic Hyrdrotherapy — FDA approved method of colon cleansing using constant warm water lavage with a contained temperature and pressure controlled device administered by a trained technician
  Other Names: Hydro San Plus Colon therapy system
  Arms: Colonic Hyrdrotherapy

SUMMARY:
The purpose of this physician blinded, randomized study is to determine the utility, effectiveness, and feasibility of using colonic irrigation as a substitute for standard oral colonic purgative solutions for colonoscopy preparation. Patients will be randomized to receive either oral isosmotic solution (PEG) or colonic irrigation using the Hydro San Plus Colon therapy system, an FDA approved and isosmotic (ISO) certified device for colonic irrigation and cleansing before endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (>18 years old) who require screening or surveillance colonoscopy
* Ability to give consent

Exclusion Criteria:

* Inability to obtain informed consent
* Pregnant patients
* Patients under the age of 18
* Active ulcerative colitis or crohn's disease flare
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of Boston Bowel Prep Score (BBPS) | 1 Day
  Quality of bowel preparations validated by numerical scale for bowel cleanse (0-9 best)

SECONDARY OUTCOMES:
Difference in Adenoma Detection Rate (ADR) | 1 Day
Difference in the number of follow ups needed after colonoscopy | 1 Day
Difference in overall comfort and convenience between Colonic Hydrotherapy and Isosmotic Irrigation using Boston Bowel Preparation Score (BBPS) | 1 Day
preferences regarding type of bowel prep for future colonoscopy based on difference in score between Colonic Hydrotherapy and Isosmotic Irrigation using Boston Bowel Preparation Score (BBPS) | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Basil Lucak, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States